CLINICAL TRIAL: NCT03018977
Title: Protocolized Sedative Weaning Versus Usual Care in Pediatric Critically Ill, Randomized Controlled Trial
Brief Title: Protocolized Sedative Weaning VS. Usual Care in Pediatric Critically Ill, RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Nattachai Anantasit, Assistant Professor, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID125808
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2017-04

CONDITIONS: Withdrawal Syndrome
MeSH Terms: conditions — Substance Withdrawal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedative weaning protocol (Active Comparator): We create the new sedative weaning protocol and then use the sedative weaning protocol.
  Interventions: Other: The sedative weaning protocol group
- Usual Care (Placebo Comparator): no use sedative weaning protocol. Sedative or/and analgesic medications are adjusted base on physician
  Interventions: Other: The usual group

INTERVENTIONS:
Other: The sedative weaning protocol group — After physician decide to wean sedative or analgesic drugs. We divided to 2 groups including high risk group and low risk group. The sedative weaning protocol were used in these patients which rely on the high risk or low risk group.
  Arms: Sedative weaning protocol
Other: The usual group — After physician decide to wean sedative or analgesic drugs. The sedative/analgesic drugs were weaned depend on physician
  Arms: Usual Care

SUMMARY:
Sedative and analgesic agents are widely used in the ICU. These agents can provide hypnotic effect, pain alleviation, cooperation, and synchronizing ventilatory support. Prolonged use of the agents can lead to withdrawal symptoms when the drugs are weaned.

Prior study showed the longer duration of sedative drugs, cumulative dose of medications and younger age were the risk factors of withdrawal syndrome. Additional, some study showed the sedation protocol can reduce the incidence of withdrawal syndrome. However, no worldwide standardized sedative weaning protocol including our hospital. The objectives in this study are to establish the sedative weaning protocol and to compare the protocol sedative weaning with the usual care weaning.

DETAILED DESCRIPTION:
Sedative and analgesic agents, particularly benzodiazepines and opioids, are widely used in PICU. These agents can provide calmness, hypnotic effect, pain alleviation, cooperation, immobilization and synchronizing ventilatory support.

Prolonged use of the agents can lead to withdrawal symptoms when the drugs are weaned.

Incidence of withdrawal syndrome is about 50%. Withdrawal syndrome can lead to unnecessary and costly diagnostic tests, prolongation of mechanical ventilation and hospital stay, and increasing of suffering. Prior study showed the longer duration of sedative drugs, cumulative dose of medications and younger age were the risk factors of withdrawal syndrome. Additional, some study showed the sedation protocol can reduce the incidence of withdrawal syndrome. However, no worldwide standardized sedative weaning protocol including our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 mo to 18 yrs, at least 37 week of postmenstrual age
* Patient who was admitted in PICU or intermediate ward at Ramathibodi hospital
* use analgesic/sedative drugs (parenteral)≥ 3 days

Exclusion Criteria:

* Patients in whom level of sedation or withdrawal assessment cannot be scored.
* Patients transferred from other hospitals in which the patients have already presented of withdrawal symptoms
* patient/parent refuse this study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01; Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
incidence of withdrawal symptom | 72 hour

SECONDARY OUTCOMES:
length of PICU stay | 30 days
sedation related adverse events | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric,Ramathibodi Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Tiacharoen D, Lertbunrian R, Veawpanich J, Suppalarkbunlue N, Anantasit N. Protocolized Sedative Weaning vs Usual Care in Pediatric Critically Ill Patients: A Pilot Randomized Controlled Trial. Indian J Crit Care Med. 2020 Jun;24(6):451-458. doi: 10.5005/jp-journals-10071-23465. PMID 32863639